CLINICAL TRIAL: NCT01106742
Title: Potential Anti-inflammatory Effect of Mushroom Extract From Agaricus Blazei Murill (ABM) in Patients With Inflammatory Bowel Disease (IBD)
Brief Title: Agaricus Blazei Murill (ABM) in Patients With Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: MD. Dag T. Førland, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbM2009-IBD
Record Dates: First submitted 2009-03-19; First posted 2010-04-20 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2009-03

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory; AbM; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — AndoSan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AndoSan, UC (Experimental): AndoSan as a supplement to 10 UC patents
  Interventions: Dietary Supplement: AndoSan
- AndoSan, CD (Experimental): AndoSan as a supplement to 10 CD patients.
  Interventions: Dietary Supplement: AndoSan

INTERVENTIONS:
Dietary Supplement: AndoSan — AndoSan, 20mlx3, 12 days
  Other Names: Agaricus blazei Murill

SUMMARY:
Based on the anti-inflammatory and stabilising effect of the AbM, (Agaricus Blazei Murill) based mushroom extract AndoSanTM on cytokine release in blood in vivo and ex vivo in healthy volunteers after 12 days consumption, the aim in this study is to investigate whether same effect is valid in patients with IBD (inflammatory bowel disease). In addition, calprotectin an abundant cytosolic protein in neutrophils and a surrogate marker for degree of intestinal inflammation will be measured in blood and feces of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderate disease activity

Exclusion Criteria:

* No use of Imurel (Azathioprin) or anti-TNF treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The ultimate goal is to see whether the ABM can be used as additional treatment of IBD. | 12 days

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Department of Surgery, Oslo, Norway